CLINICAL TRIAL: NCT04982419
Title: Remote Ischemic Preconditioning for Renal and Cardiac Protection in Congestive Heart Failure (RICH) Trial
Acronym: RICH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NEPH-019-20S; 1I01CX002045-01 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; Heart Failure; Contrast Induced Nephropathy; Coronary Angiography; Percutaneous Coronary Intervention
Keywords: Contrast-induced acute kidney injury; Congestive heart failure; Contrast induced nephropathy; Coronary angiography; Percutaneous coronary intervention; Coronary artery disease; Remote ischemic conditioning; acute coronary syndrome; Acute kidney injury; Major adverse kidney events; Ischemic preconditioning
MeSH Terms: conditions — Acute Kidney Injury; Heart Failure; Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to RIPC or sham-RIPC.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): 3 cycles of blood pressure cuff inflations to occlusive pressure of 200 mmHg for 5 minutes and deflation for 5 minutes
  Interventions: Device: Remote ischemic preconditioning
- Sham remote ischemic preconditioning (Sham Comparator): 3 cycles of blood pressure cuff inflations to non-occlusive pressure of 60 mmHg for 5 minutes and deflation for 5 minutes (Control)
  Interventions: Device: Sham remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic preconditioning — 3 cycles of blood pressure cuff inflations to occlusive pressure of 200 mmHg for 5 minutes and deflation for 5 minutes
  Other Names: RIPC
  Arms: Remote ischemic preconditioning
Device: Sham remote ischemic conditioning — 3 cycles of blood pressure cuff inflations to non-occlusive pressure of 60 mmHg for 5 minutes and deflation for 5 minutes (Control)
  Other Names: Sham-RIPC
  Arms: Sham remote ischemic preconditioning

SUMMARY:
This is a prospective, double-blind, sham-controlled, multicenter, randomized clinical trial is to study the effects of remote ischemic preconditioning on contrast-associated acute kidney injury, functional capacity, and major adverse kidney events in in patients with congestive heart failure undergoing cardiac catheterization and/or percutaneous coronary intervention.

DETAILED DESCRIPTION:
The RICH Trial is a prospective, multicenter, randomized clinical trial to determine the effect of remote ischemic preconditioning on contrast associated acute kidney injury, and to characterize the effect of remote ischemic preconditioning on brain natriuretic peptide, functional capacity at one month, and major adverse kidney events (persistent renal dysfunction, renal replacement therapy, and death) at three months in patients with congestive heart failure with reduced left ventricular ejection fraction undergoing coronary angiography and/or percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Diagnosis of heart failure with reduced LVEF <50%
* Pre-procedure intravenous normal saline fluid restriction status
* Society for Cardiovascular Angiography and Interventions (SCAI) AKI risk score (>1%)
* Referral for coronary angiogram and/or PCI
* Suspected stable coronary artery disease or acute coronary syndrome

Exclusion Criteria:

* Inability to give informed consent
* Unstable BP (SBP > 200 or <80 mmHg) at the time of enrolment
* Upper limb peripheral arterial disease
* Unavailability of at least one arm for RIPC/Sham-RIPC application
* Kidney transplant
* Renal disease requiring dialysis
* Prior exposure to contrast media within 72hrs preceding coronary angiography
* Pregnancy
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Contrast-associated acute kidney injury | 24 and 48 hours time points
  The investigators define contrast-associated acute kidney injury as a relative increase in serum creatinine of 0.3mg/dl compared with initial creatinine at 48 hours time point after coronary angiography and/or PCI. The will obtain levels of serum creatinine at baseline, then at 24 and 48 hours time points.

SECONDARY OUTCOMES:
6 minute walk distance | 1 month
  At one month follow-up, 6 minute walk test will be used to determine total distance walked in 6 minutes.
Major adverse kidney events | 3 months
  Persistent renal dysfunction, renal replacement therapy, and death will be assessed at 3 months (90 days) to determine major adverse kidney events (MAKE90).
Brain Natriuretic Peptide (BNP) | 24 and 48 hours time points
  BNP is a hormone that is primarily secreted from the ventricular myocardium in response to hemodynamic stimuli such as ventricular volume expansion and pressure overload. The investigators will obtain levels of serum BNP at baseline, then at 24 and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Oladipupo Olafiranye, MD MS, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (3):
- United States (3):
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No